CLINICAL TRIAL: NCT00195039
Title: A Phase 2 Trial of 177Lu Radiolabeled Monoclonal Antibody HuJ591-GS (177Lu-J591) in Patients With Metastatic Androgen-Independent Prostate Cancer
Brief Title: Treatment With Radiolabeled Monoclonal Antibody HuJ591-GS (177Lu-J591) in Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0304006100; 0304006100
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Results first posted 2017-10-05 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (1):
- All patients (Experimental): Eligible patients will receive a single dose of 177Lu-J591 (65 or 70 mCi/m2) consisting of J591 chelated at a specific activity of 12-15 mCi of 177Lu per mg of antibody plus sufficient non-radiolabeled, non-DOTA-conjugated ("naked") J591 to achieve a total antibody dose of 20 mg. Each dose will be administered by an IV infusion at a rate not to exceed 5 mg/min.
  Interventions: Drug: 177Lu Radiolabeled Monoclonal Antibody HuJ591 (177Lu -J591)

INTERVENTIONS:
Drug: 177Lu Radiolabeled Monoclonal Antibody HuJ591 (177Lu -J591) — Eligible patients will receive a single dose of 177Lu-J591 (65 or 70 mCi/m2) consisting of J591 chelated at a specific activity of 12-15 mCi of 177Lu per mg of antibody plus sufficient non-radiolabeled, non-DOTA-conjugated ("naked") J591 to achieve a total antibody dose of 20 mg. Each dose will be administered by an IV infusion at a rate not to exceed 5 mg/min.

SUMMARY:
The purpose of this study is to find out how effective 177Lu -J591 is in the treatment of patients with metastatic, androgen-independent prostate cancer.

DETAILED DESCRIPTION:
To determine the clinical activity of 177Lu -J591 for the treatment of patients with metastatic, androgen-independent prostate cancer.

Patients will receive a single dose of J591 (total antibody of 20 mg) consisting of antibody chelated with 177Lu at a dose of 65 or 70 mCi/m2 with a specific activity of 12-15 mCi/mg plus non-radiolabeled antibody.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of prostate adenocarcinoma.
* Metastatic prostate cancer progressive on imaging studies and/or rising PSA despite adequate medical or surgical castration therapy.
* Progressed following discontinuation of anti-androgen therapy, if received.
* Serum testosterone < 50 ng/ml

Exclusion Criteria:

* Use of corticosteroids and/or adrenal hormone inhibitors within 4 weeks of treatment.
* Use of PC-SPES within 4 weeks of treatment.
* Use of red blood cell or platelet transfusions within 4 weeks of treatment.
* Use of hematopoietic growth factors within 4 weeks of treatment.
* Prior cytotoxic chemotherapy and/or radiation therapy within 4 weeks of treatment.
* Bone scan demonstrating confluent lesions involving both axial and appendicular skeleton.
* Prior radiation therapy encompassing >25% of skeleton.
* Prior treatment with 89Strontium or 153Samarium containing compounds (e.g. Metastron®, Quadramet®).
* Active angina pectoris or NY Heart Association Class III-IV.
* History of deep vein thrombophlebitis and/or pulmonary embolus within 3 months of study entry.
* Other serious illness(es) involving the cardiac, respiratory, CNS, renal, hepatic or hematological organ systems which might preclude completion of this study or interfere with determination of causality of any adverse effects experienced in this study.
* Prior monoclonal antibody therapy with the exception of ProstaScint®
* Prior investigational therapy (medications or devices) within 6 weeks of treatment.
* Known history of HIV

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-08; Primary Completion 2012-02 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Tagawa, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medcial College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] S.T. Tagawa; M.I. Milowsky; M. J. Morris; S. Vallabhajosula; S. Goldsmith; D. Matulich; J. Kaplan; F. Berger; H. I. Scher; N. H. Bander; D. M. Nanus. Phase II trial of 177Lutetium radiolabeled anti-prostate-specific membrane antigen (PSMA) monoclonal antibody J591 in patients with metastatic castrate-resistant prostate cancer. J Clin Oncol 26: 2008 (May 20 suppl; abstr 5140)
- [Result] Tagawa ST, Milowsky MI, Morris M, Vallabhajosula S, Christos P, Akhtar NH, Osborne J, Goldsmith SJ, Larson S, Taskar NP, Scher HI, Bander NH, Nanus DM. Phase II study of Lutetium-177-labeled anti-prostate-specific membrane antigen monoclonal antibody J591 for metastatic castration-resistant prostate cancer. Clin Cancer Res. 2013 Sep 15;19(18):5182-91. doi: 10.1158/1078-0432.CCR-13-0231. Epub 2013 May 28. PMID 23714732
- [Derived] Vlachostergios PJ, Niaz MJ, Skafida M, Mosallaie SA, Thomas C, Christos PJ, Osborne JR, Molina AM, Nanus DM, Bander NH, Tagawa ST. Imaging expression of prostate-specific membrane antigen and response to PSMA-targeted beta-emitting radionuclide therapies in metastatic castration-resistant prostate cancer. Prostate. 2021 Apr;81(5):279-285. doi: 10.1002/pros.24104. Epub 2021 Jan 19. PMID 33465252

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 47
Age, Continuous [Median (Full Range); unit: years] | 73.9 [49.7 to 90.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 47
Gleason sum [Number; unit: participants] — Gleason score is the sum of 2 numbers. Primary grade is where the cancer is most prominent (or common). It is then determined where the cancer is next most prominent and assigns that region the secondary grade. A score from 1-5 is assigned for each area based on how aggressive the tumor appears. A tumor with cells that appear close to normal is assigned a low Gleason score (6 or below); low-grade tumors are less likely to spread. A tumor with cells that appear clearly different from those of a normal prostate is assigned a high Gleason score (7 or above) and is more likely to spread.
  participants
    6 | 6
    7 | 10
    8-10 | 29
    unknown | 2
PSA (ng/mL) [Median (Full Range); unit: ng/mL] | 74.4 [3.31 to 2184.6]
Sites of metastases [Count of Participants; unit: Participants]
  Bone | 46
  Lymph Node | 28
  Lung | 11
  Liver | 4
  Other | 3
ECOG performance scale [Count of Participants; unit: Participants] — 0. Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 13
    1 | 34
    2 | 0
LDH [Median (Full Range); unit: IU/L] | 217.5 [134 to 647]
Hemoglobin [Median (Full Range); unit: g/dL] | 11.9 [9.8 to 14.1]
Alkaline phosphatase [Median (Full Range); unit: IU/L] | 99 [23 to 1170]
Cancer And Leukemia Group B (CALGB) prognostic score [Median (Full Range); unit: points] — Score based on participant's Opioid analgesic use (No-Yes), LDH (</= 1xULN - >1xULN), disease site (lymph node only, bone+lymph node, any visceral), ECOG (0-2), Albumin (1-6), Hemoglobin (7-17), Alkaline Phosphatase (33-4915), PSA (0-8103.1) Once all prognostic points for predictors have been determined, the prognostic points are added for each prognostic variable. The total scale range values are 0-280. Higher values for each variable indicate earlier predicted death.
  points | 149 [88 to 184]
No. of previous hormonal therapies [Count of Participants; unit: Participants]
  1 | 6
  2 | 21
  3 | 14
  4 | 6
No. of previous chemotherapy regimens [Count of Participants; unit: Participants]
  0 | 21
  1 | 19
  >/= 2 | 7
Prior radiation [Count of Participants; unit: Participants]
  Prostate/prostate bed | 21
  Palliative to bone metastasis | 3
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Define the PSA Response Rate.
Description: PSA response rate corresponds to change form baseline in PSA at any of the time points specified.
Time Frame: At baseline, Day 1, 29, 43, 57, 85, week 18, week 24 & every 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 47
Participants
  >/= 50% decline in PSA | 5
  >/= 30% decline in PSA | 17
  Any PSA decline | 25

2. Primary Outcome: Define the Measurable Disease Response Rate.
Description: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study
Time Frame: Disease will be assessed at baseline and day 85.
Population: Only 12 patients had measurable disease
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 12
Participants
  Partial Response | 1
  Stable Disease | 8
  Progressive Disease | 2
  Lost to follow-up before repeat imaging | 1

3. Secondary Outcome: Define the Duration of Biochemical PSA and/or Measurable Disease Response.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions, Complete Response (CR) = Disappearance of all target lesions, Partial Response (PR) = A </=30% decrease in the sum of the longest diameter of target lesions, taking as reference the Baseline sum longest diameter, Stable Disease (SD) = Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter since the treatment started, Progressive Disease (PD) = A >/=20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started, or the appearance of one or more new lesions
Time Frame: At baseline, and up to death
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients
Number analyzed (Participants) | 47
months
  Any PSA decline | 22.2 [18.6 to 25.7]
  Without PSA decline | 11.4 [8.4 to 14.4]

4. Secondary Outcome: Define the Toxicity of 177Lu-J591 Given as Single Dose.
Description: Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL*.
  Grade 3 Severe or medically significant but not immediately life-threatening hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL**.
  Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: From baseline until end of treatment phase (12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 47
Participants
  Nonhematologic : ALT: Grade 1-2 | 6
  Nonhematologic : ALT: Grade 3 | 0
  Nonhematologic : ALT: Grade 4 | 0
  Nonhematologic : ALT: No toxicity | 41
  Nonhematologic : Anorexia: Grade 1-2 | 11
  Nonhematologic : Anorexia: Grade 3 | 0
  Nonhematologic : Anorexia: Grade 4 | 0
  Nonhematologic : Anorexia: No toxicity | 36
  Nonhematologic : AST: Grade 1-2 | 9
  Nonhematologic : AST: Grade 3 | 0
  Nonhematologic : AST: Grade 4 | 0
  Nonhematologic : AST: No toxicity | 38
  Nonhematologic : Bruising (no thrombocytopenia): Grade 1-2 | 2
  Nonhematologic : Bruising (no thrombocytopenia): Grade 3 | 0
  Nonhematologic : Bruising (no thrombocytopenia): Grade 4 | 0
  Nonhematologic : Bruising (no thrombocytopenia): No toxicity | 45
  Nonhematologic : Constipation: Grade 1-2 | 5
  Nonhematologic : Constipation: Grade 3 | 0
  Nonhematologic : Constipation: Grade 4 | 0
  Nonhematologic : Constipation: No toxicity | 42
  Nonhematologic : Creatinine: Grade 1-2 | 5
  Nonhematologic : Creatinine: Grade 3 | 0
  Nonhematologic : Creatinine: Grade 4 | 0
  Nonhematologic : Creatinine: No toxicity | 42
  Nonhematologic : Diarrhea: Grade 1-2 | 4
  Nonhematologic : Diarrhea: Grade 3 | 0
  Nonhematologic : Diarrhea: Grade 4 | 0
  Nonhematologic : Diarrhea: No toxicity | 43
  Nonhematologic : Dizziness: Grade 1-2 | 1
  Nonhematologic : Dizziness: Grade 3 | 0
  Nonhematologic : Dizziness: Grade 4 | 0
  Nonhematologic : Dizziness: No toxicity | 46
  Nonhematologic : Dyspepsia: Grade 1-2 | 2
  Nonhematologic : Dyspepsia: Grade 3 | 0
  Nonhematologic : Dyspepsia: Grade 4 | 0
  Nonhematologic : Dyspepsia: No toxicity | 45
  Nonhematologic : Dyspnea: Grade 1-2 | 3
  Nonhematologic : Dyspnea: Grade 3 | 0
  Nonhematologic : Dyspnea: Grade 4 | 0
  Nonhematologic : Dyspnea: No toxicity | 44
  Nonhematologic : Edema: limb: Grade 1-2 | 1
  Nonhematologic : Edema: limb: Grade 3 | 0
  Nonhematologic : Edema: limb: Grade 4 | 0
  Nonhematologic : Edema: limb: No toxicity | 46
  Nonhematologic : Fatigue: Grade 1-2 | 17
  Nonhematologic : Fatigue: Grade 3 | 0
  Nonhematologic : Fatigue: Grade 4 | 0
  Nonhematologic : Fatigue: No toxicity | 30
  Nonhematologic : Fever (without neutropenia): Grade 1-2 | 1
  Nonhematologic : Fever (without neutropenia): Grade 3 | 0
  Nonhematologic : Fever (without neutropenia): Grade 4 | 0
  Nonhematologic : Fever (without neutropenia): No toxicity | 46
  Nonhematologic : Hemorrhage, GI: oral cavity: Grade 1-2 | 1
  Nonhematologic : Hemorrhage, GI: oral cavity: Grade 3 | 0
  Nonhematologic : Hemorrhage, GI: oral cavity: Grade 4 | 0
  Nonhematologic : Hemorrhage, GI: oral cavity: No toxicity | 46
  Nonhematologic: Hypersensitivity,infusion reaction: Grade 1-2 | 11
  Nonhematologic: Hypersensitivity,infusion reaction: Grade 3 | 0
  Nonhematologic: Hypersensitivity,infusion reaction: Grade 4 | 0
  Nonhematologic: Hypersensitivity,infusion reaction: No toxicity | 36
  Nonhematologic : Nausea: Grade 1-2 | 5
  Nonhematologic : Nausea: Grade 3 | 0
  Nonhematologic : Nausea: Grade 4 | 0
  Nonhematologic : Nausea: No toxicity | 42
  Nonhematologic : Pain - abdomen NOS: Grade 1-2 | 2
  Nonhematologic : Pain - abdomen NOS: Grade 3 | 0
  Nonhematologic : Pain - abdomen NOS: Grade 4 | 0
  Nonhematologic : Pain - abdomen NOS: No toxicity | 45
  Nonhematologic : Pain - joint: Grade 1-2 | 1
  Nonhematologic : Pain - joint: Grade 3 | 0
  Nonhematologic : Pain - joint: Grade 4 | 0
  Nonhematologic : Pain - joint: No toxicity | 46
  Nonhematologic : Petechiae/purpura: Grade 1-2 | 1
  Nonhematologic : Petechiae/purpura: Grade 3 | 0
  Nonhematologic : Petechiae/purpura: Grade 4 | 0
  Nonhematologic : Petechiae/purpura: No toxicity | 46
  Nonhematologic : Rash/desquamation: Grade 1-2 | 1
  Nonhematologic : Rash/desquamation: Grade 3 | 0
  Nonhematologic : Rash/desquamation: Grade 4 | 0
  Nonhematologic : Rash/desquamation: No toxicity | 46
  Nonhematologic : Rigors/chills: Grade 1-2 | 1
  Nonhematologic : Rigors/chills: Grade 3 | 0
  Nonhematologic : Rigors/chills: Grade 4 | 0
  Nonhematologic : Rigors/chills: No toxicity | 46
  Nonhematologic : Taste alteration (dysquesia): Grade 1-2 | 1
  Nonhematologic : Taste alteration (dysquesia): Grade 3 | 0
  Nonhematologic : Taste alteration (dysquesia): Grade 4 | 0
  Nonhematologic : Taste alteration (dysquesia): No toxicity | 46
  Nonhematologic : Weight loss: Grade 1-2 | 1
  Nonhematologic : Weight loss: Grade 3 | 0
  Nonhematologic : Weight loss: Grade 4 | 0
  Nonhematologic : Weight loss: No toxicity | 46
  Hematologic : Hemoglobin: Grade 1-2 | 19
  Hematologic : Hemoglobin: Grade 3 | 5
  Hematologic : Hemoglobin: Grade 4 | 0
  Hematologic : Hemoglobin: No toxicity | 23
  Hematologic : Leukocytes (total WBC): Grade 1-2 | 14
  Hematologic : Leukocytes (total WBC): Grade 3 | 22
  Hematologic : Leukocytes (total WBC): Grade 4 | 4
  Hematologic : Leukocytes (total WBC): No toxicity | 7
  Hematologic : Neutrophils (ANC): Grade 1-2 | 7
  Hematologic : Neutrophils (ANC): Grade 3 | 17
  Hematologic : Neutrophils (ANC): Grade 4 | 12
  Hematologic : Neutrophils (ANC): No toxicity | 11
  Hematologic : Febrile neutropenia: Grade 1-2 | 0
  Hematologic : Febrile neutropenia: Grade 3 | 1
  Hematologic : Febrile neutropenia: Grade 4 | 0
  Hematologic : Febrile neutropenia: No toxicity | 46
  Hematologic : Platelets: Grade 1-2 | 4
  Hematologic : Platelets: Grade 3 | 10
  Hematologic : Platelets: Grade 4 | 22
  Hematologic : Platelets: No toxicity | 11

5. Secondary Outcome: Define the Incidence of Human Anti-J591 Antibody (HAHA) Response.
Time Frame: HAHA samples will be drawn at baseline and Day 85.
Population: Samples were collected but data necessary to summarize this outcome measure was not collected because the study team felt that there was adequate data from previous phase I studies, including repeating dosing of the study drug in this study and others that were performed prior to this study's completion.
Arm/Group | All Patients
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With Hematological Toxicity Relative to Bone Marrow Involvement (Bone Scan Index).
Description: Bone scan score determined for each patient and related to the degree of hematological toxicity quantified by % decline of nadir platelet count relative to baseline count.
Time Frame: Bone scan will be performed at baseline and Day 85.
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 47
participants | 0

7. Secondary Outcome: Assess the Survival Rate of Patients Following Treatment.
Time Frame: From baseline through study completion
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients
Number analyzed (Participants) | 47
months | 17.6 [15.2 to 20]

8. Secondary Outcome: Number of Participants With Targeting of 177Lu-J591 to Known Tumor Sites.
Time Frame: Scans will be performed between day 6 and 8.
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 47
Participants | 44

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 9/47
Other Adverse Events (participants affected / at risk) | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=47)
Bilateral Moderate Hydronephrosis (Renal and urinary disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Generalized Weakness and Fatigue (General disorders) | 1 (1)
Thrombocytopenia - grade 4 (Blood and lymphatic system disorders) | 4 (5)
Anemia - grade 3 (Blood and lymphatic system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Thrombocytopenia - grade 3 (Blood and lymphatic system disorders) | 2 (2)
Neutropenic Fever (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=47)
ALT increase (Investigations) | 6
Anorexia (Metabolism and nutrition disorders) | 11
AST increase (Investigations) | 9
Bruising (no thrombocytopenia) (Injury, poisoning and procedural complications) | 2
Constipation (Gastrointestinal disorders) | 5
Creatinine increase (Investigations) | 5
Diarrhea (Gastrointestinal disorders) | 4
Dizziness (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Edema: limb (General disorders) | 1
Fatigue (General disorders) | 17
Fever (without neutropenai) (General disorders) | 1
Hemorrhage, gastrointestinal: oral cavity (Gastrointestinal disorders) | 1
Hypersensitivity (infusion reaction) (General disorders) | 11
Nausea (Gastrointestinal disorders) | 5
Pain - abdomen NOS (General disorders) | 2
Pain - joint (General disorders) | 1
Petechiae/purpura (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Rigors/chills (General disorders) | 1
Taste alteration (dysgeusia) (Nervous system disorders) | 1
Weight loss (Investigations) | 1
Hemoglobin (Blood and lymphatic system disorders) | 24
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 40
Neutrophils (ANC) (Blood and lymphatic system disorders) | 36
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes